CLINICAL TRIAL: NCT00614367
Title: Chromosomal Analysis of Single Cells in Human Embryos
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: KU Leuven (Other)
Responsible Party: Prof Joris Vermeesch, University Hospital Leuven - Catholic University Leuven
Other Study IDs: ML4102005
Record Dates: First submitted 2008-01-30; First posted 2008-02-13 (Estimated); Last update posted 2008-02-13 (Estimated); Status verified 2008-01

CONDITIONS: Chromosomal Abnormalities
Keywords: chromosomal abnormalities in single cells
MeSH Terms: conditions — Chromosome Aberrations

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Single blastomeres of human embryos
Oversight: Data Monitoring Committee: No

SUMMARY:
Optimise genetic screening of human embryos using higher resolution techniques

ELIGIBILITY:
Inclusion Criteria:

* 3-4 day old embryos from IVF couples with both partners younger than 36 years old

Ages: 3 Days to 4 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 3-4 day old human IVF embryos
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2005-10; Primary Completion 2008-03 (Estimated); Study Completion 2008-06 (Estimated)

PRIMARY OUTCOMES:
genetic constitution of single blastomeres | 3 day old embryos

CONTACTS AND LOCATIONS:
Overall Officials: Joris Vermeesch, Prof PhD, Principal Investigator — University Hospital Leuven, Catholic University Leuven; Thomas D'hooghe, Prof MD PhD, Study Director — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospital Leuven, Catholic University Leuven, Leuven, Belgium